CLINICAL TRIAL: NCT05856773
Title: Phase III Randomized Trial of Conventionally Fractionated vs. Hypofractionated COMprehensive Nodal Irradiation for Breast Cancer Using Pencil Beam Scanning PROton Therapy (COMPRO)
Brief Title: Conventionally Fractionated vs. Hypofractionated Comprehensive Nodal Irradiation for Breast Cancer Using Pencil Beam Scanning Proton Therapy
Acronym: COMPRO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Proton Collaborative Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRE009-23
Record Dates: First submitted 2023-04-01; First posted 2023-05-12 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: Proton Radiation
MeSH Terms: conditions — Breast Neoplasms | interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A - Standard Fractionation (Active Comparator): 50-50.4 Gy (RBE) in 25-28 daily fractions of 1.8-2.0 Gy (RBE) plus a Tumor Bed Boost (for intact breast) of 10 Gy (RBE) in 4-5 daily fractions of 2-2.5 Gy (RBE)
  **Additional boost of 10-20 Gy (RBE) in 2-2.5 Gy (RBE) fractions to clinically involved lymph nodes or chest wall/scar allowed at the treating physician's discretion**
  Interventions: Radiation: Proton Therapy
- Arm B - Hypofractionation (Other): 40.05 Gy (RBE) in 15 daily fractions of 2.67 Gy (RBE) plus a Tumor Bed Boost (for intact breast) of 10 Gy (RBE) in 4-5 daily fractions of 2-2.5 Gy (RBE)
  **Additional boost of 10-20 Gy (RBE) in 2-2.5 Gy (RBE) fractions to clinically involved lymph nodes or chest wall/scar allowed at the treating physician's discretion**
  Interventions: Radiation: Proton Therapy

INTERVENTIONS:
Radiation: Proton Therapy — Pencil Beam Scanning (PBS)

SUMMARY:
The purpose of this research study is to learn more about the effects of using proton radiation therapy delivered over a shorter course of treatment (3 weeks) compared with a longer, standard course of treatment (5 weeks) for women with breast cancer who require radiotherapy to the breast/chest wall and regional lymph nodes.

DETAILED DESCRIPTION:
This study is being done to see if comprehensive regional nodal radiation therapy to the breast or chest wall and regional lymph node area using proton therapy delivered with a hypofractionated approach (less treatment days) will result in rates of treatment related skin and soft tissue side effects that are non-inferior compared to conventionally fractionated proton radiotherapy regimens.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Stage I-III breast cancer who have undergone breast conserving surgery or mastectomy and have been recommended to receive postoperative radiation therapy to the breast or chest wall and regional draining lymph nodes (axilla levels I-III, SCV, IMN)
* Histologically documented breast cancer (invasive mammary, ductal, medullary, tubular, mucinous, lobular, or ductal carcinoma in situ) for which treatment with radiation therapy to the breast/chest wall and comprehensive regional lymph nodes including the internal mammary chain is recommended
* Documentation of negative metastatic workup by whole body Positron Emission Tomography - Computed Tomography (PET/CT) or by combined CT of the chest, abdomen, pelvis and Bone scan
* History and physical exam within 90 days prior to study registration
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
* Negative pregnancy test for women of child-bearing potential
* Able to begin radiation treatment within 12 weeks of last surgery or last day of chemotherapy
* Presence of breast implants, breast expanders, tissue flap, or other breast reconstruction are allowed
* Bilateral breast cancer is allowed if at least one side will be treated with comprehensive nodal irradiation per protocol treatment and will be recorded as the laterality receiving comprehensive nodal irradiation. If both sides will be treated comprehensively, it will be documented as such

Exclusion Criteria:

* Presence of skin ulceration and / or ipsilateral satellite nodules and/or edema (including peau d'orange) (T4b or T4c disease) or diagnosis of inflammatory breast cancer (T4d disease)
* Residual gross disease detected by imaging or clinical exam with the exception of <2cm internal mammary lymph node or supraclavicular lymph node amenable to sequential boost
* Prior history of radiation therapy overlapping with current target volume (including intraoperative brachytherapy, interstitial catheter brachytherapy, balloon brachytherapy, external beam radiation therapy)
* Prior history of explant surgery or implant removal due to infection or wound healing issues without subsequent implant or flap reconstruction
* Presence of double/dual port tissue expander
* Clinical or radiographic evidence of distant metastatic disease
* Pregnant or breast-feeding females
* Non-malignant systemic disease that would preclude the patient from receiving study treatment or would prevent required follow-up
* History of connective tissue disorder (i.e., systemic lupus erythematosus, scleroderma), dermatomyositis, xeroderma pigmentosum
* Known BRCA 1 or BRCA 2 mutation
* Presence of an active skin rash
* Prior invasive non-study malignancy unless disease free for ≥ 3 years. Non-melanoma skin cancer, well-differentiated thyroid cancers, in situ carcinomas of the oral cavity, cervix, and other organs, and tumors that are not thought to impact the life expectancy of the patient are permissible.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2038-02 (Estimated); Study Completion 2041-02 (Estimated)

PRIMARY OUTCOMES:
To determine if the rate of grade ≥3 treatment-related skin and soft tissue toxicities with comprehensive nodal irradiation for breast cancer using hypofractionated PBS proton therapy is non-inferior to conventionally-fractionated proton radiotherapy | 2 years after radiation therapy
  This study will investigate if adjuvant comprehensive regional nodal radiotherapy to the breast or chest wall and regional lymph nodes including the axilla (levels I-III), supraclavicular (SCV), and internal mammary (IMN) lymph nodes using pencil beam scanning proton therapy delivered with a hypofractionated regimen results in rates of acute and late grade 3 or worse treatment-related skin and soft tissue toxicities that are non-inferior compared with rates in pencil beam scanning proton therapy using conventionally fractionated regimens.

SECONDARY OUTCOMES:
To determine the rate of any grade ≥3 treatment-related adverse events | 2, 5, and 10 years after radiation therapy
To determine local recurrence rates | 2, 5, and 10 years after radiation therapy
To determine regional recurrence rates | 2, 5, and 10 years after radiation therapy
To determine distant recurrence rates | 2, 5, and 10 years after radiation therapy
To determine breast cancer-specific survival | 2, 5, and 10 years after radiation therapy
To determine overall survival | 2, 5, and 10 years after radiation therapy
To assess patient-reported quality of life | 2, 5, and 10 years after radiation therapy
  FACT-B questionnaire
To assess patient-reported quality of life | 2, 5, and 10 years after radiation therapy
  BREAST-Q questionnaire
To assess physician-reported cosmetic outcomes | 2, 5, and 10 years after radiation therapy
  Physician reported cosmesis form

OTHER OUTCOMES:
To correlate dosimetric parameters with acute and late adverse events for the development of model dose constraints for comprehensive nodal irradiation for breast cancer using a moderately hypofractionated regimen with PBS-PT | 2, 5, and 10 years after radiation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Choi, MD, Study Chair — Proton Collaborative Group
Locations (7):
- United States (7):
  - Mayo Clinic, Scottsdale, Arizona
  - California Protons Cancer Therapy Center, San Diego, California
  - University of Florida Proton Therapy Institute, Jacksonville, Florida
  - Miami Cancer Institute, Miami, Florida
  - Emory Proton Therapy Center, Atlanta, Georgia
  - New York Proton Center, New York, New York
  - Inova Schar Cancer Institute, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No